CLINICAL TRIAL: NCT02136316
Title: A Phase 1 Study to Assess the Safety, Tolerability and Pharmacokinetics of Ascending Oral Multiple Doses of ASP7962 in Healthy Male and Female Subjects
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics (PK) of Multiple Ascending Doses of ASP7962 in Healthy Subjects
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 7962-CL-0002; 2014-000159-95 (EudraCT Number)
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Healthy Volunteers; Pharmacokinetics of ASP7962
Keywords: Healthy volunteers; ASP7962; pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ASP7962 low dose (Experimental)
  Interventions: Drug: ASP7962
- ASP7962 medium dose (Experimental)
  Interventions: Drug: ASP7962
- ASP7962 high dose (Experimental)
  Interventions: Drug: ASP7962
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASP7962 — Oral
  Arms: ASP7962 high dose; ASP7962 low dose; ASP7962 medium dose
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability as well as the pharmacokinetics of increasing oral multiple doses of ASP7962 in healthy young male and female subjects.

DETAILED DESCRIPTION:
Subjects will be admitted to the clinical unit and will stay residential for a total of 20 days/19 nights, to be discharged from the clinical unit on day 19.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index of 18.5 - 30.0 kg/m2, inclusive. Subject weighs at least 50 kg.
* Female subject must be of non-childbearing potential:

  * Postmenopausal (defined as at least 1 year without any menses and confirmation of FSH levels) prior to screening, or
  * Documented surgically sterile or status post-hysterectomy (at least 1 month prior to screening).
* Male subject and their female spouse/partner who are of childbearing potential must be using 2 highly effective forms of birth control (1 of which must be a barrier method) starting at screening and continued throughout the clinical study period, and for 90 days after the final study drug administration.
* Male subject must not donate sperm starting at screening, throughout the clinical study period, and for 90 days after the final study drug administration.
* Subject agrees not to participate in another interventional study while participating in the present clinical study, defined as signing the informed consent form until completion of the last study visit.

Exclusion Criteria:

* Subject has a known or suspected hypersensitivity to ASP7962 or any components of the formulation used.
* Subject has a history of suicide attempt or suicidal behavior. Any suicidal ideation within the last 3 months.
* Subject has any of the liver function tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase, gamma glutamyl transferase, total bilirubin [TBL]) above the upper limit of normal [ULN]. In such a case the assessment may be repeated once [day -1].
* Subject has any clinically significant history of allergic conditions.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to admission to the clinical unit on day -1.
* Subject has a mean pulse rate < 40 or > 90 bpm; mean systolic blood pressure (SBP) > 140 mmHg; mean diastolic blood pressure (DPB) > 90 mmHg (vital sign measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse rate will be measured automatically) [day -1]. If the mean pulse rate, mean SBP or mean DBP is out of the range as specified above, 1 additional triplicate measurement may be taken on day -1.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) interval > 430 ms (for male subjects) and > 450 ms (for female subjects) on admission to the clinical unit on day 1. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken [day -1].
* Subject uses any prescribed or non-prescribed drugs (including vitamins, natural and herbal remedies, e.g., St. John's wort) in the 2 weeks prior to study drug administration, except for occasional use of paracetamol (up to 2 g/day).
* Subject has used nicotine-containing products within 6 months prior to admission to the clinical unit.
* Subject has a history of drinking more than 21 units of alcohol per week for male subjects or 14 units of alcohol per week for female subjects (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months prior to admission to the clinical unit.
* Subject uses any drugs of abuse within 3 months prior to admission to the clinical unit.
* Subject uses any inducer of metabolism (e.g., barbiturates, rifampin) in the 3 months prior to admission to the clinical unit.
* Subject has had a significant blood loss, donated 1 unit (500 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to admission to the clinical unit.
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies, or antibodies to human immunodeficiency virus type 1 (HIV-1) and/or type 2 (HIV-2) at screening.
* Subject has participated in any clinical study or has been treated with any investigational drugs within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Subject is an employee of the Astellas Group or Contract Research Organization involved in the clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by adverse events | up to end of study visit (29 days)
Safety as assessed by vital signs | up to end of study visit (29 days)
Safety as assessed by orthostatic challenge test | Day 1 and 16
Safety as assessed by clinical laboratory tests | up to end of study visit (29 days)
Safety as assessed by electrocardiogram (ECG) | up to end of study visit (29 days)
  Routine 12-lead ECG, continuous cardiac monitoring (Holter ECG) and real-time cardiac monitoring (ECG telemetry)
Safety as assessed by Bond and Lader visual analogue scale (VAS) | Day 3-19
Safety as assessed by Addiction Research Center Inventory (ARCI)-49 (49-item) | Day 3-19
Safety as assessed by Columbia - Suicide Severity Rating Scale (C-SSRS) | Day 2-19
Safety as assessed by CogState cognitive test battery: Groton Maze Learning Task, Groton Maze Learning Task-Delayed Recall, Detection Task, Identification Task, One Card Learning Task, One Back Task | Day 3-19

SECONDARY OUTCOMES:
Pharmacokinetic profile of ASP7962 (plasma): AUC12, AUC12,u, AUCinf, AUCinf,u , AUClast, AUClast,u, CL/F, CLu/F, Cmax | up to Day 19
  Area under the concentration-time curve from the time of dosing to 12 hours postdose (AUC12), Area under the concentration-time curve from the time of dosing to 12 hours postdose for unbound study drug concentration (AUC12,u), Area under the concentration-time curve from time of dosing extrapolated to time infinity (AUCinf), Area under the concentration-time curve from time of dosing extrapolated to time infinity for unbound study drug concentration (AUCinf, u), Area under the concentration-time curve from the time of dosing to the last measurable concentration (AUClast), Area under the concentration-time curve from the time of dosing to the last measurable unbound concentration (AUClast, u), Apparent total systemic clearance after single or multiple extravascular dosing (CL/F), Apparent total systemic clearance of unbound study drug after single or multiple extravascular dosing (CLu/F), Maximum concentration (Cmax)
Pharmacokinetic profile of ASP7962 (plasma): Cmax,u, MRT, t1/2, tmax, tlag, λz, fu, AUCinf,u/AUCinf , Vz/F | up to Day 19
  Maximum unbound concentration (Cmax,u), Mean residence time (MRT), Terminal elimination half-life (t1/2), Time of maximum concentration (tmax), Time prior to the time corresponding to the first measurable (nonzero) concentration (tlag), Terminal elimination rate constant (λz), Fraction of study drug available systematically unbound (= free fraction) (fu), Apparent volume of distribution during the terminal elimination phase after single or multiple extravascular dosing (Vz/F)
Pharmacokinetic profile of ASP7962 (plasma): Ctrough, AUCtau, Rac(AUC), Rac(Cmax), PTR, Ratio AUCu/AUC, Vz,u/F, AUCtau,u | up to Day 19
  Concentration immediately prior to dosing at multiple dosing (Ctrough), Area under the concentration-time curve from the time of dosing to the start of the next dosing interval (AUCtau), Accumulation ratio calculated using the area under the concentration-time curve (Rac[AUC]), Accumulation ratio calculated using the maximum plasma concentration (Rac[Cmax]), Peak-trough ratio (PTR), Apparent volume of distribution during the terminal elimination phase of unbound study drug after single or multiple extravascular dosing (VZ,u/F), Area under the concentration-time curve in the dosing interval for unbound study drug concentration (AUCtau,u)
Pharmacokinetic profile of ASP7962 (urine): Aeinf, Aeinf%, Aelast, Aelast%, CLR, CLR,u, Aetau, Aetau% | Day 1 and 16
  Cumulative amount of study drug excreted into urine from time of dosing extrapolated to time infinity (Aeinf), Percentage of study drug excreted into urine from time of dosing extrapolated to time infinity (Aeinf%), Cumulative amount of study drug excreted into urine from time of dosing up to the collection time of the last measurable concentration (Aelast), Percentage of study drug excreted into urine from the time of dosing up to the collection time of the last measurable concentration (Aelast%), Renal clearance (CLR), Renal clearance of unbound study drug (CLR,u), Cumulative amount of study drug excreted into urine from the time of dosing to the start of the next dosing interval (Aetau), Percentage of study drug dose excreted into urine over the time interval between consecutive dosing (Aetau%)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Site GB44001 Parexel Early Phase Clinical Unit, London, United Kingdom